CLINICAL TRIAL: NCT01188785
Title: Phase I - Escalating Dose Study of siG12D LODER (Local Drug EluteR) in Patients With Locally Advanced Adenocarcinoma of the Pancreas, and a Single Dose Study of siG12D LODER (Local Drug EluteR) in Patients With Non-operable Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Silenseed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLSG12D
Record Dates: First submitted 2010-07-13; First posted 2010-08-25 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2014-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: siRNA; RNA interference (RNAi); Cancer; Pancreatic ductal adenocarcinoma; Pancreatic cancer; Solid tumor; Operable pancreatic ductal adenocarcinoma; Non operable pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 arm (Experimental): SOC + siG12D LODER
  Interventions: Drug: siG12D LODER

INTERVENTIONS:
Drug: siG12D LODER — Phase 0 - subjects diagnosed with an operable adenocarcinoma of the pancreas will have 8 siG12D LODER placed in tumor. The siG12D LODER will be placed in the subject's tumor using an EUS biopsy needle.
  Phase I - subjects diagnosed with locally non-operable advanced adenocarcinoma of the pancreas. These subjects will have one of three different siG12D LODERs dose levels placed in tumor - Either 1 siG12D LODER, 2 siG12D LODERs or 8 siG12D LODERs. The siG12D LODER/s will be placed in the subject's tumor using an EUS biopsy needle.

SUMMARY:
Phase 0 - Open label, Single dose study of siG12D LODER in Patients with operable adenocarcinoma of the pancreas.

The primary endpoint:

To assess efficacy and local distribution of siRNA out of eight high dose siG12D LODERs in patients diagnosed with operable adenocarcinoma of the pancreas.

The Secondary endpoint:

Short term tolerability and safety assessment

Phase I - This study is designed to investigate the safety of siG12D LODER (Local Drug EluteR) in patients diagnosed with adenocarcinoma of the pancreas.

The primary endpoint:

To asses efficacy of siG12D LODER and local distribution in non-operable patients by histopathology measurements, local distribution by RNA analysis.

To define the dose-limiting toxicities (DLT)

The Secondary endpoint

1. To determine the recommended Phase II dose (RP2D)
2. To define and maximum tolerated dose (MTD)
3. In the event of surgery, assessment of siG12D LODER local distribution and efficacy will be based on histopathology measurements and RNA analysis.
4. Progression free survival - only by long term follow-up

DETAILED DESCRIPTION:
The investigational agent siG12D LODER (Local Drug EluteR) is a miniature biodegradable polymeric matrix that encompasses anti KRASG12D siRNA (siG12D) drug, designed to release the drug regionally within a pancreatic tumor, at a prolonged rate of 12-16 weeks.

The majority of pancreatic ductal adenocarcinomas involve mutations in the KRAS oncogene (the most common is G12D), therefore stable administration of KRASG12D siRNA has the potential to silence and lead to apoptosis of such cancer cells and thereby slow and even halt the tumor growth.

ELIGIBILITY:
Inclusion Criteria:

Phase 0:

Provide written informed consent and be between the ages of 18 and up, inclusive.

* Patient that is diagnosed as respectable locally pancreatic tumor
* Have a target tumor accessible for intratumoral administration by EUS (Endoscopic Ultrasound) guidance as determined by the physician performing the EUS guided LODER insertion.
* Have a Karnofsky performance status of ≥ 70%.
* Have a life expectancy of >= 3 months.
* If female and of child-bearing potential, have a negative serum pregnancy test during screening.
* Agree to use of a barrier method of contraception if sexually active (both men and women) from the time of administration of the first treatment and for at least 8 weeks after treatment.
* Have serum creatinine < 2.0 mg/dL, , PT, - INR < 1.5 absolute neutrophil count (ANC) > 1,000 x 103 cells/mL, platelets ≥ 75,000/mL, and hemoglobin >= 10 mg/dL.
* Have screening procedures completed within 2 weeks of starting treatment.
* No other malignancy present that would interfere with the current intervention.
* Have measurable disease.

Phase I

* Provide written informed consent and be between the ages of 18 and up.
* Have an unresectable, locally advanced diagnosed or highly suspected adenocarcinoma of the pancreas. Or patients with a tumor and are not planed to undergo surgery due to a high surgical risk (e.g. coagulopathy or severe congestive heart failure).
* Allocated to receive standard of care chemo as first line treatment.
* Have a target tumor that is accessible for intratumoral administration by PTA or EUS guidance as determined by the radiologist/gastroenterologist performing the PTA/EUS injection.
* Have a Karnofsky performance status of ≥ 70%.
* Have a life expectancy of >= 3 months.
* If female and of child-bearing potential, have a negative serum pregnancy test during screening.
* Agree to use of a barrier method of contraception if sexually active (both men and women) from the time of administration of the first treatment and for at least 8 weeks after treatment.
* Have serum creatinine < 2.0 mg/dL, PT - INR < 1.5, absolute neutrophil count (ANC) > 1,000 x 103 cells/mL, platelets ≥ 75,000/mL, and hemoglobin >= 10 mg/dL.
* Have screening procedures completed within 4 weeks of starting treatment.
* No other malignancy present that would interfere with the current intervention.
* Have measurable disease.

Exclusion Criteria:

Phase 0:

* Have distant metastasis spread (such as liver or lung, or lymph nodes metastases), peritoneal spread or malignant sites.
* Have clinically significant pancreatitis within 12 weeks of treatment.
* If female, be breast feeding.
* Have a medical condition contraindicated for both percutaneous- and endoscopic- guided delivery or any intercurrent medical illness or other medical condition that would in the judgment of the investigator compromise patient safety or the objectives of the study.
* Have a history of bleeding coagulopathy.
* Have participated in any therapeutic research study within the last 4 weeks.

Phase I:

* Have distant metastatic spread (such as liver, lung, or lymph nodes metastases), peritoneal spread or malignant sites.
* Have clinically significant pancreatitis within 12 weeks of treatment.
* If female, be breast feeding.
* Have a medical condition contraindicated for both percutaneous- and endoscopic- guided delivery or any intercurrent medical illness or other medical condition that would in the judgment of the investigator compromise patient safety or the objectives of the study.
* Have a history of bleeding coagulopathy.
* Have participated in any therapeutic research study within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Phase 0 - 6 weeks, Phase I - 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Hubert, MD, Principal Investigator — Hadassah Medical Organization; Talya Golan, MD, Principal Investigator — Sheba Medical Center; Amiel Segal, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (3):
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Organization, Jerusalem
  - Sheba Medical Center, Ramat Gan

REFERENCES:
- [Derived] Golan T, Khvalevsky EZ, Hubert A, Gabai RM, Hen N, Segal A, Domb A, Harari G, David EB, Raskin S, Goldes Y, Goldin E, Eliakim R, Lahav M, Kopleman Y, Dancour A, Shemi A, Galun E. RNAi therapy targeting KRAS in combination with chemotherapy for locally advanced pancreatic cancer patients. Oncotarget. 2015 Sep 15;6(27):24560-70. doi: 10.18632/oncotarget.4183. PMID 26009994